CLINICAL TRIAL: NCT00806494
Title: A 12 Week, Multi-centre, Open Label Study To Evaluate The Efficacy, Tolerability And Safety Of A Fesoterodine Flexible Dose Regimen In Patients With Overactive Bladder.
Brief Title: UK Study Assessing Flexible Dose Fesoterodine in Adults
Acronym: SAFINA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0221058
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: Fesoterodine; Open Label; Flexible Dose; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Fesoterodine 4mg, escalating to 8mg as required
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4mg for 4 weeks, escalating to fesoterodine 8mg if tolerated

SUMMARY:
To explore the effects of fesoterodine when used in a flexible dose manner

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years old
* OAB for >3 months

Exclusion Criteria:

* Patients with conditions that would contraindicate for fesoterodine use
* Patients with significant hepatic and renal disease or other significant unstable diseases.
* OAB symptoms caused by neurological conditions, known pathologies of urinary tract, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United Kingdom (35):
  - Pfizer Investigational Site, Ely, Cambridgeshire
  - Pfizer Investigational Site, Crewe, Cheshire
  - Pfizer Investigational Site, Fowey, Cornwall
  - Pfizer Investigational Site, Penzance, Cornwall
  - Pfizer Investigational Site, Chesterfield, Derbyshire
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Baillieston, Glasgow
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Hinckley, Leicestershire
  - Pfizer Investigational Site, West Didsbury, Manchester
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Mortimer, Reading
  - Pfizer Investigational Site, Ayrshire, Scotland
  - Pfizer Investigational Site, Falkirk, Scotland
  - Pfizer Investigational Site, Winterton, Scunthorpe
  - Pfizer Investigational Site, Bath, Somerset
  - Pfizer Investigational Site, Doncaster, South Yorkshire
  - Pfizer Investigational Site, Sheffield, South Yorkshire
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, Leatherhead, Surrey
  - Pfizer Investigational Site, Worthing, West Sussex
  - Pfizer Investigational Site, Bradford-on-Avon, Wiltshire
  - Pfizer Investigational Site, Chippenham, Wilts
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Bucks
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Hertfordshire
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Northants
  - Pfizer Investigational Site, Plymouth
  - Pfizer Investigational Site, Swansea
  - Pfizer Investigational Site, Swindon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221058&StudyName=UK%20Study%20Assessing%20Flexible%20Dose%20Fesoterodine%20in%20Adults%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine: Fesoterodine 4mg tablet orally once daily (QD) for 4 weeks followed by either escalation to 8mg tablet QD or continuation of 4mg tablet QD for the remaining 8 weeks of the study treatment phase, as required.
Period: Overall Study
Arm/Group | Fesoterodine
Started | 331
Completed | 251
Not Completed | 80
Not completed — Adverse Event | 29
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 10
Not completed — Other | 30
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Fesoterodine: Fesoterodine 4mg tablet orally QD for 4 weeks followed by either escalation to 8mg tablet QD or continuation of 4mg tablet QD for the remaining 8 weeks of the study treatment phase, as required.
Arm/Group | Fesoterodine
Number analyzed (Participants) | 331
Age, Customized [Number; unit: Participants]
  Between 18 to 44 Years | 37
  Between 45 to 64 Years | 163
  >= 65 Years | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12
Description: The number of micturitions was measured by the 3-day bladder diary completed for the 3 consecutive days preceding each clinic visit. The mean number of micturitions per 24 hours was calculated as the sum of all micturitions recorded in the diary divided by the number of days the diary was completed at that visit. Change=mean at observation minus mean at baseline. Negative change, more specifically (ie), a decrease in number of micturitions relative to baseline=improvement.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS)=participants who took at least one dose of study drug and provided baseline and post-baseline data for at least 1 efficacy endpoint. N=number of participants with analyzable data. Missing data at Week 12 were imputed using last (valid post-baseline) observation carried forward (LOCF) approach.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 317
Number of Episodes | -3.26 [-3.62 to -2.91]

2. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 4
Description: The number of micturitions was measured by the 3-day bladder diary completed for the 3 consecutive days preceding each clinic visit. The mean number of micturitions per 24 hours was calculated as the sum of all micturitions recorded in the diary divided by the number of days the diary was completed at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of micturitions relative to baseline=improvement.
Time Frame: Baseline, Week 4
Population: FAS. N=number of participants with analyzable data.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 305
Number of Episodes | -2.55 [-2.87 to -2.23]

3. Secondary Outcome: Percentage Change From Baseline in the Number of Micturitions Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in micturitions was calculated as change in mean number of micturitions per 24 hours at that visit divided by the baseline mean number of micturitions per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS. n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Percentage Change
  Week 4 (n=305) | -18.69 [-20.86 to -16.51]
  Week 12 (n=317) | -23.61 [-25.86 to -21.36]

4. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturitions Per 24 Hours at Weeks 4 and 12
Description: Nocturnal micturitions were defined as those occurring between the time the subject went to bed and the time he or she arose to start the next day. The mean number of nocturnal micturitions per 24 hours was calculated as the total number of nocturnal micturitions divided by the total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of nocturnal micturitions relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (participants with nocturnal >0 micturitions per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 321
Number of episodes
  Week 4 (n=297) | -0.61 [-0.74 to -0.48]
  Week 12 (n=309) | -0.78 [-0.91 to -0.64]

5. Secondary Outcome: Percentage Change From Baseline in Nocturnal Micturitions Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in nocturnal micturitions was calculated as change in mean number of nocturnal micturitions per 24 hours at that visit divided by the baseline mean number of nocturnal micturitions per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 321
Percentage Change
  Week 4 (n=297) | -15.18 [-21.24 to -9.13]
  Week 12 (n=309) | -23.35 [-29.72 to -16.98]

6. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Weeks 4 and 12
Description: UUI episodes were defined as those with a Urinary Sensation Scale (USS) rating of 5 in the diary. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
  Mean number of UUI episodes per 24 hours was calculated as total number of micturitions with USS rating of 5 divided by total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of UUI episodes relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (number of participants with UUI episodes >0 per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 132
Number of Episodes
  Week 4 (n=125) | -1.19 [-1.52 to -0.86]
  Week 12 (n=127) | -1.64 [-2.02 to -1.25]

7. Secondary Outcome: Percentage Change From Baseline in UUI Episodes Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in UUI episodes was calculated as change in mean number of UUI episodes per 24 hours at that visit divided by the baseline mean number of episodes per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 132
Percentage Change
  Week 4 (n=125) | -59.11 [-70.61 to -47.60]
  Week 12 (n=127) | -79.30 [-88.51 to -70.10]

8. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Weeks 4 and 12
Description: Urgency episodes were defined as those with a USS rating of >=3 in the diary. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Mean number of urgency episodes per 24 hours was calculated as total number of urgency episodes divided by total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of urgency episodes relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (number of participants with urgency episodes >=3 per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Number of Episodes
  Week 4 (n=303) | -3.94 [-4.43 to -3.44]
  Week 12 (n=317) | -5.10 [-5.62 to -4.58]

9. Secondary Outcome: Percentage Change From Baseline in Urgency Episodes Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in urgency episodes was calculated as change in mean number of urgency episodes per 24 hours at that visit divided by the baseline mean number of urgency episodes per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (participants with urgency episodes >0 per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Percentage Change
  Week 4 (n=303) | -40.69 [-46.11 to -35.27]
  Week 12 (n=317) | -51.75 [-57.26 to -46.23]

10. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Urgency Episodes (NUEs) Per 24 Hours at Weeks 4 and 12
Description: NUEs were defined as those with a USS rating of >=3 in the diary, occurring between the time the participant goes to bed and the time he/she arises to start the next day. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
  Mean number of NUEs per 24 hours was calculated as total number of NUEs divided by total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of NUEs relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (participants with NUEs >0 per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 307
Number of Episodes
  Week 4 (n=284) | -0.95 [-1.10 to -0.80]
  Week 12 (n=297) | -1.16 [-1.32 to -1.01]

11. Secondary Outcome: Percentage Change From Baseline in NUEs Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in NUEs was calculated as change in mean number of NUEs per 24 hours at that visit divided by the baseline mean number of NUEs per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 307
Percentage Change
  Week 4 (n=284) | -38.71 [-45.07 to -32.35]
  Week 12 (n=297) | -44.78 [-53.41 to -36.14]

12. Secondary Outcome: Change From Baseline in Mean Number of Severe Urgency Episodes (SUEs) Per 24 Hours at Weeks 4 and 12
Description: SUEs were defined as those with a USS rating of >=4 in the diary. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine). Mean number of SUEs per 24 hours was calculated as total number of SUEs divided by total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of SUEs relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (participants with SUEs >0 per 24 hours during the 3-day baseline diary period). n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of Episodes
Arm/Group | Fesoterodine
Number analyzed (Participants) | 289
Number of Episodes
  Week 4 (n=268) | -2.31 [-2.72 to -1.90]
  Week 12 (n=278) | -2.93 [-3.36 to -2.50]

13. Secondary Outcome: Percentage Change From Baseline in SUEs Per 24 Hours at Weeks 4 and 12
Description: Percentage change from baseline in SUEs was calculated as the change in mean number of SUEs per 24 hours at that visit divided by the baseline mean number of SUEs per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; participants reporting this symptom at baseline (participants with SUEs >0 per 24 hours during the 3-day baseline diary period. n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Fesoterodine
Number analyzed (Participants) | 289
Percentage Change
  Week 4 (n=268) | -57.37 [-65.20 to -49.55]
  Week 12 (n=278) | -69.14 [-77.12 to -61.16]

14. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Pads Used Per 24 Hours at Weeks 4 and 12
Description: The mean number of incontinence pads used per 24 hours was calculated as the total number of incontinence pads used divided by the total number of diary days collected at that visit. Change=mean at observation minus mean at baseline. Negative change, ie, decrease in number of incontinence pads used relative to baseline=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS. n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Number of Incontinence Pads
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Number of Incontinence Pads
  Week 4 (n=304) | -0.49 [-0.63 to -0.35]
  Week 12 (n=316) | -0.64 [-0.79 to -0.49]

15. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Weeks 4 and 12
Description: PPBC: self-administered, single-item, questionnaire to describe perception of participants bladder-related problems (rated on 6-point scale: 1=no problems at all, 2=some very minor, 3=some minor, 4=some moderate, 5=severe, 6=many severe problems). Score change=score at observation minus score at baseline; re-scaled to 4-point categorical variables (major improvement [score difference <=-2]; minor improvement [score difference =-1]; no change [score difference = 0]; deterioration [score difference >=1]), based on PPBC score.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Number; unit: Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Participants
  Major Improvement (Week 4), n=307 | 86
  Minor Improvement (Week 4), n=307 | 121
  No Change (Week 4), n=307 | 93
  Deterioration (Week 4), n=307 | 7
  Major Improvement (Week 12), n=322 | 160
  Minor Improvement (Week 12), n=322 | 94
  No Change (Week 12), n=322 | 64
  Deterioration (Week 12), n=322 | 4

16. Secondary Outcome: Change From Baseline in Urgency Perception Scale (UPS) at Weeks 4 and 12
Description: UPS: self-administered, single-item questionnaire to measure participant's perception of urinary urgency (rated on 3-point scale: 1=usually not able to hold urine; 3=usually able to finish what I am doing before going to toilet without leaking). Score change=score at observation minus score at baseline; re-scaled to 3-point categorical variables (improvement [Increase of 1 or more points in difference of scores]; no change [score difference=0]; deterioration [Negative difference of scores], based on UPS score, with number of participants in each of the 3-point categories.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS; n=number of participants analyzed at specified timepoint. Missing data at Week 12 were imputed using LOCF approach.
Measure: Number; unit: Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Participants
  Improvement (Week 4), n=307 | 105
  No Change (Week 4), n=307 | 189
  Deterioration (Week 4), n=307 | 13
  Improvement (Week 12), n=321 | 154
  No Change (Week 12), n=321 | 159
  Deterioration (Week 12), n=321 | 8

17. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Weeks 4 and 12
Description: OAB-q symptom bother scale (8 items) is part of the OAB-q. Symptom bother score=sum of scores for items 1 to 8 (each symptom bother item measured on 6-point Likert scale ranging from 1 (not at all) to 6 (a very great deal). Lowest possible raw score=8; highest possible score=48. Data analyzed based on transformation of score to a 0 to 100 scale: (Actual total raw score - lowest possible value of raw score)/raw score range * 100. 0=no symptom bother, 100=high symptom bother. Change=mean score at observation minus mean score at baseline, negative change in score=improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS. N=number of participants with baseline score. n=number of participants analyzed at specified timepoint. Missing data at Week 12 imputed using LOCF approach.
Measure: Mean (95% Confidence Interval); unit: Score on Scale
Groups:
- Fesoteridine: Fesoterodine 4mg tablet orally once daily (QD) for 4 weeks followed by either escalation to 8mg tablet QD or continuation of 4mg tablet QD for the remaining 8 weeks of the study treatment phase, as required.
Arm/Group | Fesoteridine
Number analyzed (Participants) | 327
Score on Scale
  Week 4 (n=300) | -27.95 [-30.41 to -25.50]
  Week 12 (n=319) | -37.25 [-39.83 to -34.66]

18. Secondary Outcome: Change From Baseline in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) Score at Week 12
Description: ICIQ-SF: self-administered questionnaire for assessment and quantification of incontinence and its impact on quality of life. ICIQ score=sum of the responses to 3 questions: How often do you leak urine? (range: 0=never to 5=all the time); How much urine do you usually leak? (range: 0=none to 6=a large amount); Overall, how much does leaking urine interfere with your everyday life? (range: 0=not at all to 10=a great deal). Score range=0 (low bother from urine leakage) to 21 (maximum bother). Negative change (decrease) from baseline in score value=reduced level of bother.
Time Frame: Baseline, Week 12
Population: FAS. N=number of participants with analyzable data.
Measure: Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 305
Score on Scale | -5.13 [-5.72 to -4.54]

19. Secondary Outcome: Number of Participants With Each Categorical Response at Week 12 for Benefit, Satisfaction and Willingness to Continue (BSW) Questionnaire
Description: BSW: 3-item questionnaire to assess participants perception of effect of treatment in terms of treatment benefit, satisfaction with treatment, and participants willingness to continue treatment. Response to each item recorded in dichotomous fashion (Benefit: yes/no, yes - little benefit/much benefit; Satisfaction: yes/no, yes - a little satisfied/very satisfied, no - a little dissatisfied/very dissatisfied; Willingness to continue: yes/no, yes - a little bit willing/very willing, no - a little unwilling/very unwilling).
Time Frame: Week 12 (or Early Withdrawal)
Population: FAS, LOCF.
Measure: Number; unit: Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Participants
  Benefit from Treatment - Much Benefit | 188
  Benefit from Treatment - Little Benefit | 82
  Benefit from Treatment - No | 36
  Satisfied with Treatment - Yes | 253
  Satisfied with Treatment - No | 54
  Satisfied with Treatment - Yes (Very Satisfied) | 184
  Satisfied with Treatment - Yes (Little Satisfied) | 69
  Satisfied with Treatment - No(Little Dissatisfied) | 30
  Satisfied with Treatment - No (Very Dissatisfied) | 24
  Willingness to Continue - Yes | 248
  Willingness to Continue - No | 61
  Willingness to Continue - Yes (Very Willing) | 203
  Willingness to Continue - Yes (Little Bit Willing) | 45
  Willingness to Continue - No (Little Unwilling) | 23
  Willingness to Continue - No (Very Unwilling) | 36

20. Secondary Outcome: Percentage of Participants Reporting Satisfaction on the Treatment Satisfaction Questionnaire (TSQ) at Week 12
Description: TSQ: Independent component of the overactive bladder TSQ. Self- administered, 1-item measure of participant satisfaction for participants receiving treatment for OAB. The 5 categorical responses were grouped to 'Satisfied' (including 'very satisfied' and 'somewhat satisfied') and 'Dissatisfied' (including 'very dissatisfied','somewhat dissatisfied', and 'neither dissatisfied nor satisfied'). Percentage of participants reporting satisfaction included those with categorical responses of 'very satisfied' and 'somewhat satisfied'.
Time Frame: Week 12 (or Early Withdrawal)
Population: FAS. N=number of participants with analyzable data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 307
Percentage of Participants | 73.6

21. Secondary Outcome: Change From Baseline in King's Health Questionnaire (KHQ) Domain Scores at Week 12
Description: KHQ: Self-administered questionnaire containing 21 questions scored in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy, severity of urinary symptoms). Each domain was a categorical scale that was converted to a numeric score. All domains transformed to a range of 0 to 100, where 0=best outcome/response and 100=worst outcome/response. Change=mean score at Week 12 minus mean score at baseline, negative change from baseline=improvement.
Time Frame: Baseline, Week 12
Population: FAS. n=number of participants with analyzable data.
Measure: Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 330
Score on Scale
  General Health Perception (n=311) | -2.57 [-4.81 to -0.34]
  Incontinence Impact (n=309) | -29.69 [-32.22 to -27.17]
  Role Limitations (n=311) | -41.16 [-44.57 to -37.75]
  Physical Limitations (n=311) | -36.60 [-40.10 to -33.10]
  Social Limitations (n=310) | -25.22 [-28.38 to -22.05]
  Personal Relationships (n=220) | -15.23 [-18.77 to -11.69]
  Emotions (n=308) | -25.78 [-28.91 to -22.64]
  Sleep/Energy (n=311) | -21.38 [-24.30 to -18.47]
  Severity of Urinary Symptoms (n=311) | -21.92 [-24.49 to -19.34]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 11/331
Other Adverse Events (participants affected / at risk) | 177/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (N=331)
Angina pectoris (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Keratitis (Eye disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Oedema peripheral (General disorders) | 2
Diverticulitis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (N=331)
Dry eye (Eye disorders) | 8
Constipation (Gastrointestinal disorders) | 30
Diarrhoea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 99
Dyspepsia (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 9
Urinary tract infection (Infections and infestations) | 26
Back pain (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 7

LIMITATIONS AND CAVEATS:
This was a single arm, non-comparative study. Hence no formal hypothesis testing was performed, and assessment of efficacy was based on changes from baseline in efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.